CLINICAL TRIAL: NCT05827692
Title: UAB-CAN RULL 2022 Study: Impact of Forest Baths on Emotional Well-being in People With Sub-clinical Symptomatology of Anxiety and Depression
Brief Title: Impact of Forest Baths on Emotional Well-being in People With Sub-clinical Symptomatology of Anxiety and Depression
Acronym: NAT-UAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laura Comendador-Vazquez (Other)
Collaborators: Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor-Investigator, Laura Comendador-Vazquez, Psychologist, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022/3020
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Psychological Well-being
Keywords: forest bath; outdoor therapy; psychological well-being; RCT
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a single-center randomized controlled trial with an intrasubject pre-post design. The intervention is developed by means of two crossed treatment arms: Arm A (intervention + control); Arm B (control + intervention).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Forest Bath Intervention group A (Experimental): The intervention consists of 2 sessions of approximately 2 hours duration and fortnightly frequency. In this context, it is guaranteed that patients will receive the care, visits and treatments usually used in people who have presented their clinical situation. The only difference between participating or not in the intervention is the participation in the practice of forest baths and the performance of some additional assessments, i.e. not routinely performed, which are part of this project. The investigators will be responsible for providing an overview of the study to eligible patients interested in participating. Before proceeding to start the intervention, an informed consent will be given to the patients, in which a description of the characteristics of the sessions will be provided.
  Interventions: Behavioral: Intervention group A
- Forest Bath Intervention group B (Experimental): The intervention consists of 2 sessions of approximately 2 hours duration and fortnightly frequency. In this context, it is guaranteed that patients will receive the care, visits and treatments usually used in people who have presented their clinical situation. The only difference between participating or not in the intervention is the participation in the practice of forest baths and the performance of some additional assessments, i.e. not routinely performed, which are part of this project. The investigators will be responsible for providing an overview of the study to eligible patients interested in participating. Before proceeding to start the intervention, an informed consent will be given to the patients, in which a description of the characteristics of the sessions will be provided.
  Interventions: Behavioral: Intervention group A

INTERVENTIONS:
Behavioral: Intervention group A — The forest bath sessions will be led by a specialized guide and will be conceived as a silent walk of about 3 km along a path and forest track with an average gradient of 3%, with three 10-minute stops (at the beginning, in the middle and at the end) to practice deep breathing and awareness of the 5 senses.

SUMMARY:
The investigators intend to evaluate patients aged 18 to 99 years with symptoms of anxiety and/or mild depression. A randomized controlled clinical trial will be carried out to evaluate the impact of the guided practice of forest bathing.

DETAILED DESCRIPTION:
The practice of Shinrin-Yoku, also known as Forest Bathing, is an outdoor therapeutic modality with growing evidence suggesting positive effects on the psychological well-being and general health of individuals. However, its benefits have been studied mainly in Asian countries, needing further research to assess whether its benefits are also generalizable to other European-Mediterranean regions. To explore this question, the investigators intend to evaluate patients aged 18 to 99 years with symptoms of anxiety and/or mild depression. A randomized controlled clinical trial will be carried out to evaluate the impact of the guided practice of forest bathing. The participants will be randomly distributed in two arms, with a crossover design: arm A intervention + control; arm B control + intervention. Participation in this study consists of the execution of two sessions of guided forest bathing practice, and the completion of online evaluation forms before and after each session of guided forest bathing practice, for 24 hours afterwards, as well as before and after the program as a whole. The study includes clinical assessments, emotional well-being, social support and other complementary indicators. For hypothesis testing, a linear model of univariate analysis of variance intrasubject design will be applied to the dependent variables, with three phase conditions (pre, post and follow-up) and two treatment conditions (intervention vs. control).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 65 years.
* Voluntary signature of informed consent.
* Symptomatology of anxiety and/or mild depression with mild interference in daily functioning.
* Motivation, attitude and ability to work in a group.
* Receptive attitude to learning new skills and sharing experiences.

Exclusion Criteria:

* Serious psychiatric disorder: Major depressive disorder with or without psychotic symptoms, uncompensated major depressive episode, dysthymic disorder, presence of suicidal ideation or suicide attempts, personality disorder.
* Lack of knowledge of Catalan and Spanish.
* Disconformity with acceptable standards of conduct.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-06-18 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Generalized Anxiety Scale (GAD-7).
Change in Depression scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Patient Health Questionnaire (PHQ-9).
Change in Well-Being scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Emotional Well-Being Scale
Change in Social support scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  OSLO Scale 3
Change in State Mindfulness scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  State Mindfulness Scale (SMS)
Change in Affect scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Positive and Negative Affect Checklist (PANAS-SF).
Change in Mood scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Profile of Mood States (POMS)
Change in Stress scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Ad hoc perceived stress item
Change in Affective variables scores | Pre-intervention, intrasession, intersession, post-intervention and follo-up evaluations are planned for 1 month. The assessments will be carried out before and after the intervention with a maximum duration of 45 minutes.
  Self-Assessment Manikin (SAM)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Comendador Vázquez, Principal Investigator — Corporacion Parc Tauli
Locations (1):
- Coloma Moreno Quiroga, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No